CLINICAL TRIAL: NCT00628875
Title: "Feasibility of Ventilation Detection Using Thoracic Impedence Acquired Via Standard Defibrillator Electrode Pads in Mechanically Ventilated Pediatric Patients"
Brief Title: Feasibility of Ventilation Detection Via Standard Defibrillator Pads in Mechanically Ventilated Pediatric Patients
Acronym: Vent Detection
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Laerdal Medical (Industry)
Responsible Party: Kathryn Roberts, Children's Hospital of Philadelphia
Other Study IDs: 2006-10-5022
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: Respiration, Artificial
Keywords: mechanical ventilation; thoracic impedence; defibrillator pads; ventilation detection; pediatric ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a prospective, observational case series of a convenience sample of mechanically ventilated pediatric patients in the Pediatric ICU, Progressive Care Unit and Operating Room at the Children's Hospital of Philadelphia.

We propose to observe, measure and report the accuracy, precision and bias of defibrillator electrode pads to detect breathing in stable but critically ill and mechanically ventilated children. This study will provide preliminary data to inform the resuscitation research community and assist development of evidence-based pediatric resuscitation guidelines in the future.

DETAILED DESCRIPTION:
Context: Resuscitation (CPR) guidelines recommend target values for rate and depth of rescue breathing and chest compressions. Defibrillator electrode pads can accurately detect the size, rate, and speed of machine-generated breaths in adults. The accuracy, precision, bias, and ability of the defibrillator electrode pads to detect the size, rate and speed of breathing in children have not been studied.

Objectives: The primary objective is to evaluate the accuracy, precision, bias and ability of the pads and defibrillator to detect the rate and depth of breathing in critically ill children on breathing machines. Important secondary objectives include reporting the accuracy, precision and bias of the measurement of the speed of the breath, measurement variability, and impact of alternative defibrillator electrode pad location on the chest.

Study Design/Setting/Participants:

Prospective, pilot, observational study in the Pediatric Intensive Care Unit and Progressive Care Unit at the Children's Hospital of Philadelphia. The participants are all patients in the PICU and Progressive Care Unit (PCU), 6 months to 17 years, who are supported by their clinical management team with a tracheal tube, standard breathing machine, and standard ICU monitoring systems.

Intervention:

Standard defibrillator electrode pads will be placed on the patient's chest in two typical pediatric configurations, and data will be recorded for 5 minutes in each configuration. These defibrillator electrode pads will be used exclusively for monitoring, as additions to the standard ICU monitoring.

Study Measures:

The primary outcome variable will be the successful detection of breathing rate. We will compare the accuracy, precision and bias of detection of each breath of > 2 ml/kg by the defibrillator electrode pads compared with the "gold standard" mechanical ventilator pneumotachometer detected breaths. Secondary outcome variables will include defibrillator electrode pad detection of breathing depth and speed compared to standard ICU monitors (considered the gold standard). We will also study the effect of defibrillator electrode pad location on the accuracy, precision, bias and ability to detect breathing rate, depth, and speed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 6 months - 17 years with:
2. Artificial airway
3. Mechanical ventilation (PCV or VCV)
4. Hemodynamic stability to participate in the study, as determined by the clinical treatment team.
5. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Patients with chest tubes
2. High frequency ventilation (Jet or Oscillation)
3. Airway Pressure Release ventilation
4. Extracorporeal membrane oxygenation (ECMO)
5. Significant chest wall abnormality (e.g. Vertebral Expandable Prosthetic Titanium Rib (VEPTR) or device precluding typical placement of defibrillator electrode pads)
6. Altered skin integrity in areas where defibrillator electrode pads would be placed

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients admitted to the Pediatric Intensive care Unit, Progressive Care Unit or Operating Room at the Children's Hospital of Philadelphia
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
This is a pilot study to gather preliminary data. The primary endpoint is the accuracy of defibrillator pad detection of breaths >2ml/kg, compared to the gold standard pneumotachometer detection of breaths. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Roberts, MSN, RN, CRNP, CCRN, CCNS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States